CLINICAL TRIAL: NCT06650202
Title: Improving Balance After Spinal Cord Injury Using a Robotic Upright Stand Trainer and Spinal Cord Epidural Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Gail Forrest, Associate Director, Tim and Caroline Reynolds Center for Spinal Stimulation, Kessler Foundation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R-1243-23
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-10

CONDITIONS: SCI - Spinal Cord Injury
Keywords: TPAD
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: A total of 20 spinal cord injured participants who were previously implanted with a spinal cord epidural stimulation (scES) unit will be enrolled and split into two groups with 10 participants in each. All participants will undergo a physical examination and classification of their spinal cord injury to determine eligibility criteria, which are the same for both groups. Participants will then be placed into one of the two groups based on their availability and preference. Group 1 will consist of individuals with SCI and an scES implant that will receive TPAD training with stimulation and assessments with and without stimulation. Group 2 will consist of individuals with SCI and an scES implant that will only receive assessments with and without stimulation. Each participant will serve as their own control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1- Training and Assessments (Other): 10 SCI participants with an scES implant that will receive 40-60 TPAD training sessions with stimulation and 5 assessments with and without stimulation.
  Interventions: Device: The Tethered Pelvic Assist Device (TPAD)
- Group 2- Assessments Only (No Intervention): 10 SCI participants with an scES implant that will receive 4 assessments with and without stimulation.

INTERVENTIONS:
Device: The Tethered Pelvic Assist Device (TPAD) — a light-weight cable-driven robotic stand trainer that (i) can provide assistance-as-needed by applying corrective forces on the trunk and pelvis in response to their movement outside a pre-programmed area, and (ii) can apply controlled forces on the trunk and pelvis to perturb them from their nominal configuration during standing.
  Arms: Group 1- Training and Assessments

SUMMARY:
The purpose of this study is to understand how standing and sitting balance control is altered after spinal cord injury and how a new type of robotic assistive device may be used with spinal stimulation to improve muscle function. The investigators will be testing a device called the Tethered Pelvic Asist Device (or "TPAD") in this study. The TPAD may be helpful in two ways. It can be used to help control and support of the trunk, pelvis, and knees during stand training. Also, the TPAD can be used as a training tool by providing controlled "pushes" or "perturbations" that must be corrected by the person with spinal cord injury in order to maintain proper posture and upright balance. This could be helpful for improving muscle function after spinal cord injury.

Participants will be placed into one of two groups based on availability and preference. Group 1 will receive TPAD training with stimulation and assessments with and without stimulation. Participation in this group lasts approximately 4 months. Group 2 will only receive assessments with and without stimulation. Participation in this group last approximately 3 weeks.

DETAILED DESCRIPTION:
The aims of the proposed study are to (a) examine the muscle activation patterns generated during stable and perturbed standing in spinal cord injured individuals using spinal cord epidural stimulation (scES) and robotic TPAD-assistance or self-assistance for balance, and (b and c) to examine the effectiveness of TPAD-assisted stand training in the improvement of postural control during stable and perturbed standing and sitting in spinal cord injured individuals using spinal cord epidural stimulation (scES).

The Tethered Pelvic Assist Device (TPAD) is a light-weight cable-driven robotic stand trainer that (i) can provide assistance-as-needed by applying corrective forces on the trunk and pelvis in response to their movement outside a pre-programmed area, and (ii) can apply controlled forces on the trunk and pelvis to perturb them from their nominal configuration during standing.

A total of 20 spinal cord injured participants who were previously implanted with a scES unit will be enrolled in this study. They will be split into two groups with 10 participants in each. All participants will undergo a physical examination and classification of their spinal cord injury to determine eligibility criteria, which are the same for both groups. Participants will then be placed into one of the two groups based on their availability and preference to be enrolled in a longer or shorter study. Group 1 will consist of individuals with SCI and an scES implant that will receive TPAD training with stimulation and assessments with and without stimulation. Group 2 will consist of individuals with SCI and an scES implant that will only receive assessments with and without stimulation.

Each individual will serve as their own control, to reduce variability. All participants will undergo the Stable Standing Assessment, Postural Perturbation Assessment, Stable Sitting Assessment and Postural Perturbation Assessment in Sitting. Only Group 1 will also perform the Neuromuscular Recovery Scale and attend training sessions with the TPAD system.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Stable medical condition.
* Has a spinal cord injury caused by trauma (fall, car accident, etc.) for at least one year that is not getting worse over time
* Has an implanted spinal cord epidural stimulation unit that is eligible for software upgrade as part of a previous study.
* Unable to stand independently with epidural stimulation turned off.

Exclusion Criteria:

* unwilling to discontinue from anti-spasticity medications
* Untreated painful problems with joints, muscles or bones.
* Unhealed fracture.
* Pressure sore or urinary tract infection.
* History of bone disease (except for decreased bone mineral density due to spinal cord injury).
* Ongoing drug abuse.
* Untreated psychiatric disorders or clinical depression.
* Received Botox injections in the lower extremities in the prior six months.
* Heart or lung disease that may interfere with assessments.
* Untreated severe and persistent problems regulating blood pressure, heart rate, body temperature or other automatic functions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Neuromuscular Recovery Scale (NRS) | On average, 2 hours to complete. Group 1will complete the NRS at the beginning of the study and at the end (on average 4 months)
  Research participants will undergo a series of tasks to test the level of muscle activation and amount of assistance required during standing and stepping in a body-weight supported treadmill environment, as well as overground motor tasks. Arm, trunk/leg movement recovery and independency will be measured by the NRS using 14 motor tasks (sit, reverse sit up, sit up, sitting truck extension, overhead press, forward reach and grasp, door pull and open, can open and manipulation, sit to stand, stand, walking, stand adaptability, step retraining, and step adaptability) and combined with EMG, kinematic, and kinetic analyses on the upper and lower extremities and/or trunk. Based on the performance across categories, 4 phase scores can be assigned:1- greatest impairment relative to normal movement patterns (non-ambulatory), 2- begins to stand and weight support independently, 3- walking with varying skill levels, and 4- normal locomotor and transfer performance with adaptability.
Sitting Assessment | On average 4 hours to complete. Done at the beginning and end of the study by both groups (group 1: 4 months, group 2: 3 weeks). Repeated by group 1 during training up to 4 times.
  Research participants will sit on a padded table and perform tasks to challenge their balance control (reaching/shifting weight in multiple directions). Assistance for sitting will be provided at the trunk by the TPAD or by the trainer. EMG and kinematic analysis will be performed on the lower extremities, trunk and upper extremities during sitting. The trunk force and position controller data from the TPAD will be also collected; these data will be synchronized with EMG and kinematic data. Muscle activation patterns will be evaluated recording EMG from different muscle groups. The TPAD/trainer will then generate controlled loss of balance during sitting. EMG onset and burst duration relative to perturbation onset, loss of balance onset and return to balance will be compared. EMG mean and integrated amplitudes from each muscle will be compared between the beginning and end of the study.
Standing Assessment | On average 4 hours to complete. Done at the beginning and end of the study by both groups (group 1: 4 months, group 2: 3 weeks). Repeated by group 1 during training up to 4 times.
  Participants will stand as long as possible and undergo a series of standing tasks. Electromyography (EMG), kinematic and kinetic analysis will be performed on the lower extremities and trunk during standing. The pelvic, trunk and knee force and position controller data from the TPAD will be collected and synchronized. Muscle activation patterns will be evaluated recording EMG from different muscle groupings. When appropriate, ground reaction forces will be measured. Blood pressure and heart rate will be measured. The TPAD will then generate controlled loss of balance during standing. Participants will regain balance with/without grasping a fixed object. Investigators will compare EMG onset and burst duration relative to perturbation onset, loss of balance onset and return to balance if applicable. EMG mean and amplitudes from each muscle will be compared before and after the study.

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
All Individual Participant Data (IPD) will be kept with the study research team at Kessler Foundation. IPD will be de-identified and may be shared with the device research team at Columbia University, the FDA, Kessler Foundation Institutional Review Board, the Department of Health and Human Services, and collaborators at the Kentucky Spinal Cord Injury Research Center.